CLINICAL TRIAL: NCT01395537
Title: Phase I/II Pilot Study of Lapatinib in Combination With Carboplatin and Paclitaxel in the Treatment of Recurrent/Metastatic Adenocarcinoma of the Esophagus and Gastroesophageal Junction (GEJ)
Brief Title: Lapatinib With Carboplatin and Paclitaxel in Esophagus and Gastroesophageal Junction (GEJ)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Research Cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2310
Record Dates: First submitted 2011-07-12; First posted 2011-07-15 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Paclitaxel; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib With Carboplatin and Paclitaxel (Experimental)
  Interventions: Drug: Carboplatin AUC; Drug: Paclitaxel; Drug: lapatinib

INTERVENTIONS:
Drug: Carboplatin AUC — Carboplatin AUC 6 IV over 30 minutes on day one of a three week cycle. This will be continued for 6 cycles or until progression of disease or intolerable side effects.
Drug: Paclitaxel — Paclitaxel 175 mg/m2 IV over 3 hours day one of a three week cycle. This will be continued for 6 cycles or until progression of disease or intolerable side effects.
Drug: lapatinib — Lapatinib should be taken once daily, at the same time daily, on an empty stomach, either 1 hour before, or 1 hour after meals.

SUMMARY:
RATIONALE: Since lapatinib inhibits both EGFR and HER2 receptors, it is an attractive agent for the treatment of esophageal and GEJ tumors.

PURPOSE: Lapatinib is currently approved for HER2 positive metastatic breast cancer in combination with capecitabine or letrozole. It is hoped that by giving lapatinib and carboplatin and paclitaxel together, their combined effects will further slow or stop the cancer cells from growing.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Phase I: To assess the toxicity and feasibility of the addition of lapatinib to carboplatin and paclitaxel in patients with recurrent/metastatic adenocarcinoma of the esophagus and gastroesophageal junction.
2. Phase II: To assess the response rate to this regimen.

OUTLINE:

1. There will be an initial phase I safety cohort studies requiring up to 12 patients, followed by a phase II cohort using the lapatinib dose defined in phase I. Carboplatin and paclitaxel doses will not be escalated.

   The initial dose of lapatinib of 750 mg daily by mouth will be given to 6 patients. There will be no dose escalation of the lapatinib above 1000 mg daily. The lapatinib dose for the phase II cohort of this trial will be based only on toxicities experienced during the first cycle (3 weeks) of treatment.
2. Phase II: Once the optimal lapatinib dose has been chosen, all remaining patients will initiate treatment at this dose level. Patients with stable or responding disease after 6 cycles will continue treatment with lapatinib alone until progression of disease or intolerable side effects. Feasibility, toxicity and response rate of this combination will be assessed.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of adenocarcinoma of the esophagus, or gastroesophageal junction based on biopsy material or adequate cytologic exam.
* Patients must have incurable metastatic or recurrent adenocarcinoma of esophagus or gastroesophageal junction.
* Patients must have an ECOG performance status of 0-1.
* Patients must have adequate bone marrow function as evidence by: absolute neutrophil count > 1500/uL, and platelet count > 100,000/uL
* Patients must have adequate renal function as evidenced by a Cockcroft-Gault calculated creatinine clearance > 30 mL/min.
* Patient must have adequate hepatic function as evidenced by: serum total bilirubin < 2.0 mg/dl, and AST/ALT < 3 X the institutional upper limit of normal. Patients with an elevated unconjugated bilirubin (Gilbert's syndrome) will be eligible if hepatic enzymes and function are otherwise completely normal (AST/ALT/Alk Phos within normal limits), and there is no evidence of hemolysis.
* Patients must have cardiac ejection fraction > 50% as measured by echocardiogram or MUGA scan.
* Patient must agree to stop medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of lapatinib. (See Appendix I).
* Patients must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must have measurable/evaluable disease as per RECIST 1.1 criteria.
* Tumor must be tested for HER2 and EGFR before patient registration.
* Patients of childbearing potential must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method).
* Patients must be >18 years old.
* Women of childbearing potential must have a negative pregnancy test prior to enrollment.
* Patients must have a life expectancy >12 weeks.
* Patients must be able to tolerate oral (or feeding-tube administered) medications.

Exclusion Criteria:

* Patients with any other diagnosis except for adenocarcinoma (squamous cell carcinoma, small cell carcinoma, lymphoma, etc) will be ineligible.
* Patients with another active malignancy within the last 5 years will not be eligible except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with PSA <1.0 mg/dL on 2 successive evaluations at least 3 months apart, with the most recent evaluation within 4 weeks of entry.
* Patients may not have had any previous chemotherapy for recurrent or metastatic disease and no chemotherapy or radiation therapy within the past 4 weeks.
* Patients may not have received any previous treatment with carboplatin, paclitaxel, or a HER2 or EGFR inhibitor prior to enrollment.
* Patients may not be receiving any other investigational agents or other concurrent anticancer therapy.
* Patients with brain metastases are excluded.
* Patients with > grade 2 peripheral neuropathy per NCI's Common Toxicity Criteria Version 4.0 will be ineligible.
* Males with QTc > 450 or females with QTc > 470msec will be ineligible.
* Patients with active cardiac disease are excluded including current uncontrolled or symptomatic angina, history of clinically significant arrhythmias requiring medications, (with the exception of asymptomatic atrial tachycardias requiring anticoagulation and/or beta-blockade), myocardial infarction < 6 months from study entry, uncontrolled or symptomatic congestive heart failure, or any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Women who are currently pregnant or lactating will be ineligible.
* Any other uncontrolled inter-current medical or psychiatric illness.
* Known HIV-positive patients will be excluded.
* Patients with any gastrointestinal disease resulting in an inability to take oral )or feeding-tube administered medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Adelstein, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Neelesh Sharma, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from medical clinic from 8/2011 to 4/2013.
Period: Phase I
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
Started | 13
Completed | 13
Not Completed | 0
Period: Phase II
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
Started (Only one participant was eligible to move to the phase II part of the study.) | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 58 [43 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: PHASE I: Number of Patients That Experience a Grade 3-4 Dose Limiting Toxicity
Description: A dose limiting toxicity (DLT) will be defined as any grade 3-4 non-hematologic toxicity or increase in bilirubin >/= 2 mg/dL (>2X baseline in patients with Gilbert's syndrome), or elevation in AST/ALT > 3.0 X ULN during the first 3 week course of therapy.
Time Frame: after 9 weeks (3 cycles) of treatment
Population: All participants that received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
Number analyzed (Participants) | 13
Participants | 1

2. Primary Outcome: PHASE II: To Assess the Response Rate to This Regimen.
Description: Number of patients with stable or responding disease after 6 cycles of carboplatin and paclitaxel will continue treatment with lapatinib alone until progression of disease or intolerable side effects.
Time Frame: after 37 months
Population: Participants eligible to move to phase II of study. Study was cancelled prior to additional participants moving to study.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: To Determine the Overall Survival
Description: Overall survival is defined as the length of time between the date of starting treatment and death due to any cause. For a patient who is alive at the time of the statistical analysis, the patient will be considered censored at the last date of known contact.
Time Frame: after 37 months
Population: Participants that received treatment
Measure: Median (Full Range); unit: weeks
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
Number analyzed (Participants) | 13
weeks | 32 [15 to 75]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while participants were on study ranging from 4 to 19 months.
Arm/Group | Lapatinib With Carboplatin and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 13/13
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib With Carboplatin and Paclitaxel (N=13)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib With Carboplatin and Paclitaxel (N=13)
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1 (2)
anemia (Blood and lymphatic system disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 7 (10)
dysphagia (Gastrointestinal disorders) | 6 (8)
fatigue (General disorders) | 2 (4)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
infusion reaction (General disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (2)
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 6 (6)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (1)
Neutropenia (Investigations) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
peripheral neuropathy (Nervous system disorders) | 1 (3)
platelets, decreased (Investigations) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
rash on nose and chin (Skin and subcutaneous tissue disorders) | 1 (1)
right upper quadrant pain (Gastrointestinal disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
weight loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
One patient was treated in phase II cohort. The study was then prematurely terminated because of the results of the TRIO-013/LOGiC trial. It failed to meet its primary survival endpoint, suggesting little justification for continuation of our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes